CLINICAL TRIAL: NCT01440959
Title: A Phase II Trial of TKI258 in Patients With Metastatic or Advanced Gastrointestinal Stromal Tumors (GIST) After Failure to Imatinib and Sunitinib(CTKI258AKR01T)
Brief Title: Dovitinib for Imatinib/Sumitinib-failed Gastrointestinal Stromal Tumors (GIST): TKI258
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Study Principal Investigator, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC1403
Record Dates: First submitted 2011-09-08; First posted 2011-09-27 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: This is a single-center; prospective; single-arm; open-label phase II study
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TKI258 (Experimental)
  Interventions: Drug: dovitinib

INTERVENTIONS:
Drug: dovitinib — TKI258 at 500 mg/day on a 5 days on/2 days off dosing schedule
  Other Names: A phase II study of TKI258

SUMMARY:
With discovery of KIT mutations and the advent of KIT tyrosine kinase inhibitor imatinib (GlivecTM, Novartis), there has been substantial improvement in overall survival in patients with advanced and/or metastatic gastrointestinal tumors (GIST). Recently, sunitinib (SuteneTM, Pfizer) showed activity as second-line therapy in GIST patients after failure with imatinib. However, virtually all patients will eventually progress or become intolerable after the first-line imatinib and the second-line sunitinib. Dovitinib (TKI258, Novartis) is a multi-kinase inhibitor. TKI258 is a potent inhibitor of the VEGFR 1, 2, and 3, FGFR1, 2 and 3, PDGFRβ, Kit, RET, TrkA, CSF 1R, and FLT3 with inhibitory concentration 50% (IC50s) of less than 40nM. Stem cell factor (SCF) also termed KIT ligand, or steel factor has been shown to modulate tumor angiogenesis. In cultured human endothelial cells and Kit expressing cancer cells, TKI258 inhibits VEGF- and SCF-stimulated mitogenesis. .

DETAILED DESCRIPTION:
It is well known that KIT and PDGFR which can be inhibited by TKI258 have a crucial role in the development and proliferation of GIST, and in general FGFR has an important role in angiogenesis and tumor proliferation in many cancers. We assume that TKI258 can be also effective in patients with GIST. The objective of this study is to evaluate the safety and activity of TKI258 given as salvage treatment for GIST after failure to standard imatinib and sunitinib.

ELIGIBILITY:
Inclusion criteria

* Age 20 years or older
* Histologically confirmed metastatic and/or advanced GIST with CD117(+), DOG-1(+), or mutation in KIT or PDGFRα gene
* Failed (progressed and/or intolerable) after prior treatments for GIST, including at least both imatinib and sunitinib .
* ECOG performance status of 0~2
* Resolution of all toxic effects of prior treatments to grade 0 or 1 by NCI-CTCAE version 3.0
* At least one measurable lesion as defined by RECIST version 1.0.
* Adequate bone marrow, hepatic, renal, and other organ functions

  * Neutrophil > 1,500/mm3
  * Platelet > 75,000/mm3
  * Hemoglobin > 8.0 g/dL
  * Total bilirubin < 1.5 x upper limit of normal (ULN)
  * AST/ALT < 2.5 x ULN (or < 5 x ULM in case of liver metastases)
  * Creatinine < 1.5 x ULN
  * Amylase, lipase < ULN
* Electrolytes should be within normal limits.
* Urine dipstick reading: Negative for proteinuria or, if documentation of +1 results for protein on dipstick reading, then total urinary protein ≤ 500 mg and measured creatinine clearance ≥ 50 mL/min/1.73m2 from a 24-hour urine collection
* Life expectancy > 12 weeks
* Women with reproductive potential must have a negative serum or urine pregnancy test
* Washout period of previous TKIs or chemotherapy for more than 4 times the half life.
* Provision of a signed written informed consent

Exclusion criteria

* Women of child-bearing potential who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control.
* Clinically significant cardiac disease (New York Heart Association, Class III or IV) or impaired cardiac function or clinically significant cardiac diseases,
* Uncontrolled infection.
* Diabetes mellitus (insulin dependent or independent disease, requiring chronic medication) with signs of clinically significant peripheral vascular disease.
* Previous pericarditis; clinically significant pleural effusion in the previous months or current ascites requiring two or more interventions/month.
* Known pre-existing clinically significant disorder of the hypothalamic-pituitary axis, adrenal or thyroid glands.
* Prior acute or chronic pancreatitis of any etiology.
* Acute and chronic liver disease and all chronic liver impairment.
* Malabsorption syndrome or uncontrolled gastrointestinal toxicities with toxicity greater than NCI CTCAE grade 2.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality.
* Treatment with any of the medications that have a potential risk of prolonging the QT interval or inducing Torsades de Points and the treatment cannot be discontinued or switched to a different medication prior to starting study drug.
* Use of ketoconazole, erythromycin, carbamazepine, phenobarbital, rifampin, phenytoin and quinidine 2 weeks prior baseline.
* Major surgery ≤ 28 days prior to starting study drug or who have not recovered from side effects of such therapy.
* Known diagnosis of HIV infection .
* History of another primary malignancy that is currently clinically significant or currently requires active intervention.
* Patients with brain metastases as assessed by radiologic imaging
* Alcohol or substance abuse disorder.
* no other inhibitor of FGFR except sunitinib

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2011 and April 2012, a total of 30 patients with metastatic and/or unresectable GISTs who had treatment failure with imatinib and sunitinib were enroled in Asan Medical Center, Seoul, Korea.
Pre-assignment Details: There are no specific approaches between enrollment and treatment.
Groups:
- TKI258: dovitinib : TKI258 at 500 mg/day on a 5 days on/2 days off dosing schedule
Period: Overall Study
Arm/Group | TKI258
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TKI258
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 30

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR; OR + Stable Disease)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR; Progressive disease (PD), >20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD), Insufficient change to qualify for PR or PD
  This was evaluated with abdominal and pelvic dynamic CT scan every 4 weeks for the initial 8 weeks, and then every 8 weeks.
Time Frame: Up to 24 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TKI258
Number analyzed (Participants) | 30
Percentage of participants | 13 [4.7 to 30.3]

2. Secondary Outcome: Overall Response Rate Using Both CT and PET Scans
Description: PET scan will be performed at baseline and at 4 weeks of treatment. Metabolic response was defined based on the PET response criteria of the European Organization for Research and Treatment of Cancer (EORTC); a metabolic partial response (mPR) was defined as a 25% reduction in average SUVmax; metabolic stable disease (mSD) between a 25% decrease and 25% increase in average SUVmax; metabolic progressive disease (mPD) as a 25% increase in average SUVmax or the appearance of new uptake in metastatic lesions.
Time Frame: Up to 24 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | TKI258
Number analyzed (Participants) | 30
Percentage of participants
  Response rate by CT | 3
  Response rate by PET | 13

3. Secondary Outcome: Efficacy According to the Primary Mutation Type
Description: Correlation between efficacy results such as response, progression-free survival and overall survival, and primary mutation type including KIT exons 9, 11, 13, and 17 and PDGFRα exons 12 and 18.
Time Frame: Up to 24weeks
Reporting Status: Not Posted

4. Secondary Outcome: Efficacy According to the Concentrations of Circulating Growth Factors
Description: Correlation between efficacy results, such as response, progression-free survival, and overall survival andcirculating growth factors (including vascular endothelial growth factor, fibroblast growth factor, interleukin-8, placental growth factor, and fibroblast growth factor23), and soluble receptors (including soluble form of membrane bound vascular endothelial growth factor receptor-1 and -2).
Time Frame: Up to 24weeks
Reporting Status: Not Posted

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be graded according to Common Terminology Criteria for Adverse events version 3.0, up to 3 year.
Time Frame: Monitoring of adverse events will be continued for at least 28 days following the last dose of study treatment, up to 3 year.
Measure: Number; unit: participants
Arm/Group | TKI258
Number analyzed (Participants) | 30
participants | 30

6. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from the first treatment to the onset of progressive disease per RECIST criteria or to the date of death whichever comes first. For patients who do not experience progressive disease or death, the progression-free survival duration will be right censored on the last disease assessment date.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TKI258
Number analyzed (Participants) | 30
months | 3.6 [3.5 to 3.7]

7. Secondary Outcome: Overall Survival
Description: Overall survival duration is calculated as time from the first treatment to the date of death. For patients who are still alive at the cut-off date for statistical reporting, the overall survival duration will be right censored on the last known alive date.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TKI258
Number analyzed (Participants) | 30
months | 9.7 [6.0 to 13.4]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | TKI258
Serious Adverse Events (participants affected / at risk) | 8/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TKI258 (N=30)
Anorexia (Gastrointestinal disorders) | 1 — Grade 2 anorexia
Left ventricular systolic dysfunction (Cardiac disorders) | 1 — Grade 3 heart failure
QT prolongation (Cardiac disorders) | 1 — grade 4 QT prolongation
Plumonary thromboembolism (Cardiac disorders) | 1 — Grade 3 pulmonary thromboembolism
Thrombocytopenia (Blood and lymphatic system disorders) | 2 — Grade 3 thrombocytopenia
Azotemia (Renal and urinary disorders) | 1 — grade 2 azotemia
Cataract (Eye disorders) | 1 — Grade 3 cataract
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TKI258 (N=30)
Neutropenia (Blood and lymphatic system disorders) | 11
Anemia (Blood and lymphatic system disorders) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Anorexia (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 19
Asthenia (General disorders) | 18
Hypertension (Cardiac disorders) | 13
Proteinuria (Renal and urinary disorders) | 10
Skin rash (Skin and subcutaneous tissue disorders) | 9
Headache (Nervous system disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 12
Azotemia (Renal and urinary disorders) | 18
Elevated aspartate aminotransferase (Hepatobiliary disorders) | 12
Elevated alanine transaminase (Hepatobiliary disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No